CLINICAL TRIAL: NCT06540573
Title: The Relationship Between Serum Chemokine Ligand 21 (CCL-21) Level and Disease Activity in Patients With Rheumatoid Arthritis and Osteoarthritis
Brief Title: The Relationship Between Serum Chemokine Ligand 21 (CCL-21) Level and Disease Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 450
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
Keywords: C-C Motif Chemokine Ligand 21; Rheumatoid Arthritis; Osteoarthritis; Disease severity
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients who were diagnosed with osteoarthritis and applied to outpatient clinic: Patients diagnosed with osteoarthritis (meeting the American College of Rheumatology (ACR) criteria
  Interventions: Diagnostic Test: Laboratory tests (examination); Diagnostic Test: Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index; Diagnostic Test: Patient global assessment (PGA); Diagnostic Test: Physician global assessment (PhGA); Diagnostic Test: Health Assessment Questionnaire (HAQ); Diagnostic Test: Knee Radiography
- Patients who were diagnosed with rheumatoid arthritis and applied to outpatient clinic: Patients diagnosed with rheumatoid arthritis (meeting the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 criteria
  Interventions: Diagnostic Test: Laboratory tests (examination); Diagnostic Test: The Disease Activity Score28 (DAS28); Diagnostic Test: Patient global assessment (PGA); Diagnostic Test: Physician global assessment (PhGA); Diagnostic Test: Health Assessment Questionnaire (HAQ); Diagnostic Test: Clinical disease activity index (CDAI); Diagnostic Test: The Simplified Disease Activity Index (SDAI)
- Healthy volunteers: Healthy who were volunteers applied to the physical treatment and rehabilitation outpatient clinic
  Interventions: Diagnostic Test: Laboratory tests (examination); Diagnostic Test: Health Assessment Questionnaire (HAQ)

INTERVENTIONS:
Diagnostic Test: Laboratory tests (examination) — Laboratory tests (examination) to be performed include complete blood count, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), liver function tests and kidney function tests; rheumatoid factor (RF), anti-cyclic citrullinated peptide antibody (anti-CCP antibody) and C-C Motif Chemokine Ligand 21 (CCL21).
Diagnostic Test: Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index — Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) This questionnaire is used to assess the health status of osteoarthritis patients introduced in 1988 (13). It is consisted of 33 items which evaluates the health and function of the patient from various aspects including: clinical symptoms (5 questions), severity of joint stiffness (2 questions), degree of pain (9 questions), and activity of daily living (17 questions).The test questions are scored on a scale of 0-4, which correspond to: None(0),Mild (1),Moderate (2),Severe(3),and Extreme (4).The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores.Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
  Groups: Patients who were diagnosed with osteoarthritis and applied to outpatient clinic
Diagnostic Test: The Disease Activity Score28 (DAS28) — The Disease Activity Score (DAS) was created as a numerical tool for quantifying and assessing disease activity in rheumatoid arthritis (RA).The DAS28 (Disease Activity Score using 28 joint counts) was developed from the original DAS (Disease Activity Score).The DAS28 evaluates the disease activity by assessing the number of tender and swollen joints in a patient. Specifically, it considers 28 joints. The DAS28 also takes into account a blood marker of inflammation, typically the erythrocyte sedimentation rate (ESR) or the C-reactive protein (CRP) level.A patient with a DAS28 score of less than 2.6 is in remission; a score greater than or equal to 2.6 and less than 3.1 indicates low activity; a score greater than or equal to 3.1 and <5.1 indicates moderate activity and a score 5.1 or more indicates high activity
  Groups: Patients who were diagnosed with rheumatoid arthritis and applied to outpatient clinic
Diagnostic Test: Patient global assessment (PGA) — Patient global assessment (PGA) of disease activity will be reported by patients. PGA was developed in the late 1970s and was initially designed for the measurement of self-assessed pain in RA [8], although it has since been used to evaluate RA more globally. It is interesting to note that the way PGA is used in clinical practice covers, in fact, two very different concepts, one related to global health and the other to overall disease activity. They are both usually used under the heading of PGA without further specification for which is being assessed.
  Groups: Patients who were diagnosed with osteoarthritis and applied to outpatient clinic; Patients who were diagnosed with rheumatoid arthritis and applied to outpatient clinic
Diagnostic Test: Physician global assessment (PhGA) — Physician global assessment (PhGA)of disease activity will be reported by the physician.The Physician Global Assessment (PhGA) of treatment response measures the overall response to treatment as assessed by the physician. The PhGA is a well accepted and commonly used scale for evaluating treatment response in clinical trials both in adults and children. PhGA is a simple instrument and the result is easily understood. However, assigning a score for PhGA requires a very detailed evaluation. To perform this assessment a physician/health care provider would use extensive data from every aspect of ICF.
  Groups: Patients who were diagnosed with osteoarthritis and applied to outpatient clinic; Patients who were diagnosed with rheumatoid arthritis and applied to outpatient clinic
Diagnostic Test: Health Assessment Questionnaire (HAQ) — Functional impairment will be assessed with the Health Assessment Questionnaire (HAQ). It is a self-assessment tool used to measure functional ability in eight different areas: rising, dressing and grooming, hygiene, eating, walking, reach, grip, and activities of independent living. Each item or question is rated on a scale of 0 to 3, with 0 (normal/no difficulty), 1 (some difficulty), 2 (much difficulty), and 3 (unable to do). The 8 category scores are averaged, which represent an overall score from 0 (no disability) to 3 (completely disabled). If the questionnaire is slightly changed to reflect a certain disease, this does not affect the respective scoring.Scores 0-1 indicates mild to moderate disability, 1-2 indicates moderate to severe disability, and 2-3 indicates severe to very severe disability.
Diagnostic Test: Clinical disease activity index (CDAI) — Clinical Disease Activity Index (CDAI) is a composite index (without acute-phase reactant) for assessing disease activity. CDAI is based on the simple summation of the count of swollen/tender joint count of 28 joints along with patient and physician global assessment on VAS (0-10 cm) Scale for estimating disease activity. The CDAI has range from 0 to 76
  Groups: Patients who were diagnosed with rheumatoid arthritis and applied to outpatient clinic
Diagnostic Test: The Simplified Disease Activity Index (SDAI) — The Simplified Disease Activity Index for Rheumatoid Arthritis (SDAI) is a scoring system that has been validated in both research and clinical settings. It has been shown to have the highest sensitivity and specificity for predicting a physicians' decisions to change DMARD therapy when compared to other scores.Remission is defined as an SDAI of <3.3, low disease activity as ≤11, moderate disease activity as ≤26 and high disease activity as >26. Response to therapy is considered moderate if SDAI decreases by ≥7 and major if decreases by ≥17
  Groups: Patients who were diagnosed with rheumatoid arthritis and applied to outpatient clinic
Diagnostic Test: Knee Radiography — Knee osteoarthritis (gonarthrosis) will be evaluated using Kellgren-Lawrence (KL) staging on direct radiographs (anteroposterior and lateral views).Numerous variations of the Kellgren and Lawrence classification system have been used in research. Grade 0 (none): definite absence of x-ray changes of osteoarthritis. Grade 1 (doubtful): doubtful joint space narrowing and possible osteophytic lipping.Grade 2 (minimal): definite osteophytes and possible joint space narrowing. Grade 3 (moderate): moderate multiple osteophytes, definite narrowing of joint space, some sclerosis and possible deformity of bone ends Grade 4 (severe): large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends. Osteoarthritis is deemed present at grade 2 although of minimal severity
  Groups: Patients who were diagnosed with osteoarthritis and applied to outpatient clinic

SUMMARY:
Rheumatoid arthritis (RA) is a chronic systemic disease characterized by the development of new capillaries involved in the infiltration of inflammatory cells causing synovial hyperplasia and progressive destruction of cartilage and bone.Osteoarthritis (OA) is a degenerative joint disease that involves articular cartilage and other intra-articular structures.Although the pathological mechanisms involved in OA and RA are different, the onset and progression of both diseases are associated with inflammation, immune mechanisms and metabolic factors.C-C Motif Chemokine Ligand 21 (CCL21) is a CCR7-binding chemokine that plays an important role by modulating the circulation of T cells and dendritic cells in lymphoid and peripheral organs (9). Ligation of CCL21 in RA fibroblasts and macrophages induced the production of proangiogenic factors such as VEGF, Ang-1, and IL-8, suggesting that CCL21 plays an indirect role in RA angiogenesis.The aim of our study is to evaluate the serum levels of CCL21 in RA and OA patients by comparing them with healthy controls. In addition, the aim is to examine the correlation of serum CCL21 with disease degree/severity in both diseases and to determine whether it can be a biomarker of the disease state.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic systemic disease characterized by the development of new capillaries involved in the infiltration of inflammatory cells causing synovial hyperplasia and progressive destruction of cartilage and bone. The synovial tissue layer consists of macrophages and fibroblasts, which have profound effects on the destructive process in RA through the production of pro-inflammatory cytokines, chemokines and pro-angiogenic factors (2,3). Osteoarthritis (OA) is a degenerative joint disease that involves articular cartilage and other intra-articular structures (4). OA leads to pain, stiffness, decreased joint function (5), and ultimately disability (6). Although the pathological mechanisms involved in OA and RA are different, the onset and progression of both diseases are associated with inflammation, immune mechanisms and metabolic factors (7,8). C-C Motif Chemokine Ligand 21 (CCL21) is a CCR7-binding chemokine that plays an important role by modulating the circulation of T cells and dendritic cells in lymphoid and peripheral organs (9). Ligation of CCL21 in RA fibroblasts and macrophages induced the production of proangiogenic factors such as VEGF, Ang-1, and IL-8, suggesting that CCL21 plays an indirect role in RA angiogenesis ( 10 ).

We determined that CCL21-mediated RA arthritis extends joint inflammation to bone erosion by coupling the differentiation of M1 macrophages with Th17 cells. Disease progression is further exacerbated by CCL21-induced neovascularization. We conclude that CCL21 is an attractive new target for the treatment of RA, as blocking its function can abolish erosive arthritis modulated by M1 macrophages and Th17 cell crosstalk. In short, CCL21 is a pleiotropic chemokine that shapes many aspects of RA pathology. We have not found a study that examined CCL21 blood serum levels in RA and OA patients and healthy controls and evaluated whether there is a relationship between CCL21 and these diseases.

The aim of our study is to evaluate the serum levels of CCL21 in RA and OA patients by comparing them with healthy controls. In addition, the aim is to examine the correlation of serum CCL21 with disease degree/severity in both diseases and to determine whether it can be a biomarker of the disease state.

ELIGIBILITY:
Inclusion Criteria:

* 20 RA patients, 20 Osteoarthritis patients and 20 healthy volunteers between the ages of 16-60.

Exclusion Criteria:

* Age < 16 years,
* Systemic Disorders (Diabetes, Hematological diseases (coagulopathies), serious cardiovascular diseases, chronic liver and kidney disease or malignancy.)
* Patients suffering from infectious disorders (septic arthritis, viral arthritis, fungal arthritis and other rheumatic diseases such as spondyloarthropathies, systemic lupus erythematosus or dermatomyositis and others.)
* Individuals with other autoimmune diseases, malignancy, cardiac or neurological deficits, end-stage organ failure and other conditions that may affect the serum level of CCL21, such as diabetes mellitus, concomitant inflammatory disease (acute infection or chronic inflammatory state), coronary artery disease and hepatitis, were excluded from the study. was left
* Lymphadenopathies
* OA patients who received intra-articular injection or systemic glucocorticoid therapy within 3 months were excluded from the study.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Selection of all patient and healthy control volunteers was carried out at Gaziosmanpasa Training and Research Hospital Physical Medicine and Rehabilitation Department; It was conducted consecutively from rheumatology outpatient clinics. 20 healthy volunteers, 20 patients diagnosed with Osteoarthritis (meeting the American College of Rheumatology (ACR) criteria), and 20 patients diagnosed with Rheumatoid Arthritis (meeting the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 criteria) will be included in the study. Written and verbal consent will be obtained from all individuals included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The Disease Activity Score28 (DAS28) | Within 1 week of applying to outpatient clinic
  The Disease Activity Score (DAS) was created as a numerical tool for quantifying and assessing disease activity in rheumatoid arthritis (RA).The DAS28 (Disease Activity Score using 28 joint counts) was developed from the original DAS (Disease Activity Score).The DAS28 evaluates the disease activity by assessing the number of tender and swollen joints in a patient. Specifically, it considers 28 joints. The DAS28 also takes into account a blood marker of inflammation, typically the erythrocyte sedimentation rate (ESR) or the C-reactive protein (CRP) level.A patient with a DAS28 score of less than 2.6 is in remission; a score greater than or equal to 2.6 and less than 3.1 indicates low activity; a score greater than or equal to 3.1 and <5.1 indicates moderate activity and a score 5.1 or more indicates high activity
Patient global assessment (PGA) | Within 1 week of applying to outpatient clinic
  Patient global assessment (PGA) of disease activity will be reported by patients. PGA was developed in the late 1970s and was initially designed for the measurement of self-assessed pain in RA [8], although it has since been used to evaluate RA more globally. It is interesting to note that the way PGA is used in clinical practice covers, in fact, two very different concepts, one related to global health and the other to overall disease activity. They are both usually used under the heading of PGA without further specification for which is being assessed.
Physician global assessment (PhGA) | Within 1 week of applying to outpatient clinic
  Physician global assessment (PhGA)of disease activity will be reported by the physician.The Physician Global Assessment (PhGA) of treatment response measures the overall response to treatment as assessed by the physician. The PhGA is a well accepted and commonly used scale for evaluating treatment response in clinical trials both in adults and children. PhGA is a simple instrument and the result is easily understood. However, assigning a score for PhGA requires a very detailed evaluation. To perform this assessment a physician/health care provider would use extensive data from every aspect of ICF.
Health Assessment Questionnaire (HAQ) | Within 1 week of applying to outpatient clinic
  Functional impairment will be assessed with the Health Assessment Questionnaire (HAQ). It is a self-assessment tool used to measure functional ability in eight different areas: rising, dressing and grooming, hygiene, eating, walking, reach, grip, and activities of independent living. Each item or question is rated on a scale of 0 to 3, with 0 (normal/no difficulty), 1 (some difficulty), 2 (much difficulty), and 3 (unable to do). The 8 category scores are averaged, which represent an overall score from 0 (no disability) to 3 (completely disabled). If the questionnaire is slightly changed to reflect a certain disease, this does not affect the respective scoring.Scores 0-1 indicates mild to moderate disability, 1-2 indicates moderate to severe disability, and 2-3 indicates severe to very severe disability.
Clinical disease activity index (CDAI) | Within 1 week of applying to outpatient clinic
  Clinical Disease Activity Index (CDAI) is a composite index (without acute-phase reactant) for assessing disease activity. CDAI is based on the simple summation of the count of swollen/tender joint count of 28 joints along with patient and physician global assessment on VAS (0-10 cm) Scale for estimating disease activity. The CDAI has range from 0 to 76
Simplified Disease Activity Index | Within 1 week of applying to outpatient clinic
  The Simplified Disease Activity Index for Rheumatoid Arthritis (SDAI) is a scoring system that has been validated in both research and clinical settings. It has been shown to have the highest sensitivity and specificity for predicting a physicians' decisions to change DMARD therapy when compared to other scores.Remission is defined as an SDAI of <3.3, low disease activity as ≤11, moderate disease activity as ≤26 and high disease activity as >26. Response to therapy is considered moderate if SDAI decreases by ≥7 and major if decreases by ≥17

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Dag, Study Chair — Eyup Sultan State Hospital

REFERENCES:
- [Result] Li G, Zhao J, Li B, Ma J, Zhao Q, Wang X, Lv Z, Li K, Du Z, Ma X, Liu J. Associations between CCL21 gene polymorphisms and susceptibility to rheumatoid arthritis: a meta-analysis. Rheumatol Int. 2017 Oct;37(10):1673-1681. doi: 10.1007/s00296-017-3784-4. Epub 2017 Aug 10. PMID 28799100
- [Result] Van Raemdonck K, Umar S, Palasiewicz K, Volkov S, Volin MV, Arami S, Chang HJ, Zanotti B, Sweiss N, Shahrara S. CCL21/CCR7 signaling in macrophages promotes joint inflammation and Th17-mediated osteoclast formation in rheumatoid arthritis. Cell Mol Life Sci. 2020 Apr;77(7):1387-1399. doi: 10.1007/s00018-019-03235-w. Epub 2019 Jul 24. PMID 31342120